CLINICAL TRIAL: NCT06029166
Title: Electrocardiographic Changes and Rhythm Disorders Associated With BTK Inhibitors Exposure Using an Insertable Subcutaneous Cardiac Monitor: a Multicenter Cardio-Oncology Prospective Cohort
Brief Title: Subcutaneous Cardiac Monitoring of Patients With BTK Inhibitors
Acronym: IRAF-ISCM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Collaborators: University Hospital, Marseille (Other); Groupe Hospitalier Pitie-Salpetriere (Other); European Georges Pompidou Hospital (Other); Hôpital Necker-Enfants Malades (Other); Saint Antoine University Hospital (Other); Hospices Civils de Lyon (Other); Centre Hospitalier Universitaire de Saint Etienne (Other); Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 22-0252
Record Dates: First submitted 2023-08-28; First posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-07

CONDITIONS: Atrial Fibrillation
Keywords: cardio-oncology; cardiotoxicity; hematologic malignancy; atrial fibrillation; rhythm disorders; insertable subcutaneous cardiac monitor
MeSH Terms: conditions — Atrial Fibrillation; Cardiotoxicity; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hematologic malignancy patients requiring a treatment by Bruton's tyrosine kinase inhibitor (Other): Consecutive adult patients with a definite diagnosis of hematologic malignancy requiring a treatment by Bruton's tyrosine kinase (BTK) inhibitor (ibrutinib, acalabrutinib, zanubrutinib) during at least 12 months will be included to receive an insertable subcutaneous cardiac monitor (ISCM).
  Interventions: Device: Insertable subcutaneous cardiac monitor (BIOMONITOR IIIm®, Biotronik®)

INTERVENTIONS:
Device: Insertable subcutaneous cardiac monitor (BIOMONITOR IIIm®, Biotronik®) — Implantation of a subcutaneous cardiac monitor (BIOMONITOR IIIm®, Biotronik®) before beginning the Bruton's tyrosine kinase inhibitor treatment.

SUMMARY:
The goal of this clinical trial is to screen all types of electrocardiographic changes and rhythm disorders in adult patients with a hematologic malignancy requiring a treatment by Bruton's tyrosine kinase (BTK) inhibitor (ibrutinib, acalabrutinib, zanubrutinib) using an insertable subcutaneous cardiac monitor (ISCM) and occurring from inclusion and within 12 months.

This study consists of the implantation of an ISCM at inclusion and before BTK inhibitor initiation. Then patients will have medical visits every 3 months (+/- 7 days) during 12 months and a continuous cardiac telemonitoring using the ISCM.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients,
* Definite diagnosis of hematologic malignancy requiring a BTK inhibition with ibrutinib, acalabrutinib or zanubrutinib,
* Expected BTK inhibitor duration estimated to be at least 12 months,
* Sinus rhythm at enrolment,
* Willing to sign patient consent form and to comply with scheduled visits, as outlined in the protocol

Exclusion Criteria:

* Age < 18 years old,
* Adults with protective measures (curatorship or tutorship) and vulnerable patients,
* Pregnant or nursing women,
* Permanent atrial fibrillation or long-standing persistent atrial fibrillation as defined by the European Society of Cardiology guidelines,
* Atrial fibrillation on the electrocardiogram at the inclusion visit,
* Previous left atrial ablation or previous maze or maze-like surgery,
* Indication for or patients with a pacemaker or implantable cardioverter-defibrillator at baseline,
* Untreated hyperthyroidism,
* Uncorrected kaliaemia disorders at the inclusion visit,
* Hemoglobin < 8 g/L at the inclusion visit,
* Thrombopenia < 50,000/mm3 at the inclusion visit,
* Active bleeding,
* Myocardial infarction < 1 month,
* Surgery < 1 month,
* Mechanical heart valve,
* Valvular heart disease requiring surgery,
* Inability to follow the required procedures of the clinical investigation plan,
* No signature of patient consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of any electrocardiographic changes and/or rhythm disorders from first BTK inhibitors prescription to 12 months of follow-up, symptomatic or not, detected on 12-lead ECG and/or on ISCM. | 3, 6, 9 and 12 months after introduction of ibrutinib therapy (+/- 7 days)
  Electrocardiographic changes and/or rhythm disorders are defined by the European Society of Cardiology guidelines.

SECONDARY OUTCOMES:
Electrocardiographic intervals (PR, QRS, QT) measurements on both 12-lead ECG and ISCM at baseline and with BTK inhibitors exposure. | 3, 6, 9 and 12 months after introduction of ibrutinib therapy (+/- 7 days)
The occurrence of bleeding events from inclusion and within 12 months. | 3, 6, 9 and 12 months after introduction of ibrutinib therapy (+/- 7 days)
Correlation between IRAF and multiple demographic, clinical, cardiac imaging (morphological data) and serum cardiac biomarkers. | 3, 6, 9 and 12 months after introduction of ibrutinib therapy (+/- 7 days)
IRAF management. | 3, 6, 9 and 12 months after introduction of ibrutinib therapy (+/- 7 days)
Progression-free survival of patients treated by BTK inhibitors according to the presence of IRAF. | 3, 6, 9 and 12 months after introduction of ibrutinib therapy (+/- 7 days)
Correlation between QT/QTc measurements performed by ISCM (BIOMONITOR IIIm®, Biotronik®) and a QT expert on 12-leads ECG. | 3, 6, 9 and 12 months after introduction of ibrutinib therapy (+/- 7 days)
Daily body temperature monitoring with the ISCM (BIOMONITOR IIIm®, Biotronik®) temperature sensor and will be compared with conventional body temperature measurements performed during follow-up visits. | 3, 6, 9 and 12 months after introduction of ibrutinib therapy (+/- 7 days)
Constitute a plasmatic biobank for futures ancillary studies. | 3, 6, 9 and 12 months after introduction of ibrutinib therapy (+/- 7 days)
The need for ISCM (BIOMONITOR IIIm®, Biotronik®) remove within the 12-months follow-up. | 3, 6, 9 and 12 months after introduction of ibrutinib therapy (+/- 7 days)

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Department of Pharmacology, Caen, Normandy, France

IPD SHARING:
Plan to Share IPD: Undecided